CLINICAL TRIAL: NCT06283108
Title: The Impact of Distraction During Transition to the Operating Room and Anesthesia Induction Using a Novel Virtual Reality Software Program on Pediatric Perioperative Anxiolysis and Induction Compliance.
Brief Title: Gurney Journey: Virtual Reality Distraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Colorado (Other)
Responsible Party: Principal Investigator, Aline Maddux, Physician, Critical Care, Children's Hospital Colorado
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-1183
Record Dates: First submitted 2024-02-22; First posted 2024-02-28 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Dental Caries in Children; Dental Diseases; Gastrointestinal Surgery; Procedures Requiring Anesthesia
Keywords: pediatric; induction
MeSH Terms: conditions — Stomatognathic Diseases | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Virtual Reality Experimental (Experimental): Standard CCLS care and distraction with Virtual Reality
  Interventions: Device: Standard Child Life Preparation and Support + Meta Quest 2 VR headset with Gurney Journey (a mixed reality experience)
- Standard CCLS care (Active Comparator): Standard CCLS care
  Interventions: Behavioral: Standard Child Life Preparation and Support

INTERVENTIONS:
Device: Standard Child Life Preparation and Support + Meta Quest 2 VR headset with Gurney Journey (a mixed reality experience) — Certified Child Life Specialist's will provide preparation and support for patients before and during their anesthesia induction for their dental or gastrointestinal procedure. Child life specialist's will utilize Gurney Journey as part of their support for induction. Gurney Journey is a mixed reality experience, using the Meta Quest 2 VR headset that was designed to mitigate patient anxiety during transport from pre-admission rooms to the procedure room/operating room for surgical procedures.
  Arms: Virtual Reality Experimental
Behavioral: Standard Child Life Preparation and Support — Certified Child Life Specialist's will provide preparation and support for patients before and during their anesthesia induction for their dental procedure.
  Arms: Standard CCLS care

SUMMARY:
The aim of this study is to determine whether a software virtual reality (VR) program provided during transportation to anesthesia induction reduces anxiety before the procedure, and compliance in pediatric patients. This study aims to measure the anxiety of patients as they arrive before their procedure, when parting from their parents for transportation to the procedure room, and when anesthesia is provided. Compliance during anesthesia induction will also be monitored. Participants will be randomly placed into to one of two groups. Group 1 will receive standard care from a Certified Child Life Specialist prior to their surgery. Group 2 will receive standard care from a Certified Child Life Specialist and distraction with a novel virtual reality software program.

DETAILED DESCRIPTION:
The aim of this study is to determine whether a novel software virtual reality (VR) program provided during transition from periop to the procedure room and anesthesia induction reduces preoperative anxiety, and induction compliance in pediatric patients. This study aims to specifically monitor and measure the anxiety of patients as they arrive at the preoperative suite, when parting from their parents for transportation to the procedure room, and at induction of anesthesia. Compliance during anesthesia induction will also be monitored. Participants will be randomized to one of two groups. Group 1 will receive standard care during their surgery. Group 2 will receive standard care and distraction with a novel virtual reality software program. We hypothesize that anxiety will be reduced, and anesthesia compliance will improve for participants in Group 2.

ELIGIBILITY:
Inclusion Criteria:

* Ages 5-17 years old.
* Patients undergoing general anesthesia with mask induction for dental or gastrointestinal procedures.

Exclusion Criteria:

* Cognitive impairment that will impact the use of the VR headset or interaction with the game.
* Participants who cannot comfortably wear the VR headset.
* Visual impairment that would hinder use of software program.
* Patients receiving general anesthesia via IV.
* Parent accompanies patient back for anesthesia induction.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2024-04-19 (Actual); Primary Completion 2025-06-03 (Actual); Study Completion 2025-06-03 (Actual)

PRIMARY OUTCOMES:
modified Yale Preoperative Anxiety Scale | Perioperative, transport to operating room, in operating room
  Observational scale used to measure patient anxiety at different time points. Higher scores mean the patient is displaying more anxiety. Scores range from 23.33 to 100.
Induction Compliance Checklist | In operating room at induction
  Used to measure and observe a patient's compliance with anesthesia induction. It uses a checklist of 10 items that correspond to negative behaviors that are frequently observed at such time, scoring 1 point for each measure on the checklist. The score is obtained by summing the scores for all the items (10 points maximum). Perfect anesthetic induction (with no negative behaviors) scores 0 points, suboptimal induction is scored between 1 and 4 and a score above 4 is considered as poor induction.

SECONDARY OUTCOMES:
The Pediatric Behavioral Induction Assessment | After induction
  Measure completed by anesthesiologist's in the procedure room to describe patients' behavior during induction of anesthesia.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No